CLINICAL TRIAL: NCT02124057
Title: Evaluation of Hepatic Function in Patients With Spinal and Bulbar Muscular Atrophy
Brief Title: Study of Hepatic Function in Patients With Spinal and Bulbar Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140099; 14-N-0099
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Spinal and Bulbar Muscular Atrophy (SBMA); Motor Neuron Disease
Keywords: Liver; Motor Neuron Disease; Natural History
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (5):
- Healthy female control: Age-matched healthy control women
- Healthy male control: Age-matched healthy control men
- Other Motor Neuron Disease Patients: Male participants with other motor neuron disease
- SBMA Patients: Men with genetically confirmed SBMA
- SMBA: SBMA carrier women

SUMMARY:
Background:

- Spinal and bulbar muscular atrophy (SBMA) is an inherited disease. It causes weakness in muscles used for swallowing, breathing, and speaking. SBMA mainly affects men, but women can carry the gene for it. Researchers think there may be a link between SBMA and excess fat in the liver.

Objective:

- To look for fatty liver and liver injury in people with SBMA, people with motor neuron disease, and people who carry the gene for SBMA.

Eligibility:

* Adults 18 years and older who have SBMA, have motor neuron disease, or are carriers of SBMA.
* Healthy adult volunteers.

Design:

* Participants will be screened with medical history, physical exam, and blood tests.
* Participants will have 1 outpatient visit of 1-2 days. Women will have a urine pregnancy test. All participants will have:
* Blood tests.
* Liver ultrasound. A probe is placed on the abdomen at certain locations and angles and takes pictures. The painless procedure takes 20-30 minutes.
* Liver magnetic resonance imaging (MRI) scan. The MRI scanner is a metal cylinder with a magnetic field. Participants will lie on a table that slides in and out of it. They will be in the scanner for about 30 minutes. They will get earplugs for loud noises.
* Some participants with abnormal liver testing will have a biopsy (small piece) of the liver taken. The biopsy site will be located with ultrasound, then cleaned and numbed. The physician will quickly pass a needle in and out of the liver while the participants holds their breath. Afterward, participants will be monitored in bed for 6 hours.
* Participants may return for follow-up and another 1-2 day outpatient visit yearly for up to 2 years.

DETAILED DESCRIPTION:
Objectives:

Spinal and bulbar muscular atrophy (SBMA), or Kennedy s disease, is a slowly progressive hereditary motor neuron disease for which there is currently no effective treatment. Whether the liver is affected in SBMA is unclear. Preliminary analysis in SBMA patients has shown changes including increased hepatic fat, which requires additional investigation. Female carriers and patients with motor neuron disease will also participate in the study to evaluate for liver fat and function via imaging and laboratory tests.

Study Population:

We plan to enroll 15 men with genetically confirmed SBMA, 15 age-matched healthy control men, 15 SBMA carrier women, 15 age-matched healthy control women and 15 males with other motor neuron disease patients as disease controls. As of September 2017, recruitment is complete for men with genetically confirmed SBMA (n=15 recruited), age-matched healthy control men (n=15 recruited), SBMA carrier women (n=14 recruited), and 15 age-matched healthy control women (n=14 recruited). Recruitment of motor neuron disease subjects as disease controls for the study began in April 2018 and is ongoing. Our goal is to recruit 12 more disease control subjects.

Design:

Subjects will complete liver evaluations at the NIH that may include blood work, liver MRI imaging with spectroscopy (MRS), ultrasound, and biopsy. Liver biopsy will be performed on a subset of subjects with SBMA only, who have a clinical indication for biopsy analysis. Liver tissue will be analyzed by the NIH Clinical Center Pathology Department, and additional studies will be done in the research laboratory at NIH. Patients may undergo repeated non-invasive testing to determine if the liver findings are changing over time. An evaluation of muscle fat by MRI spectroscopy will be done with a subset of up to 10 subjects receiving the liver studies.

Outcome measures:

Subjects will be assessed using several different types of measurements including blood work for fatty metabolism, muscle function, and hepatic function. Liver biopsies will be used to determine the pattern and degree of fatty infiltration in SBMA patients. Liver and muscle imaging will be used to detect fat. Ultrasound elastography will be used to assess the extent of fibrosis and loss of elasticity in the liver.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study population will consist of several subgroups of patients. An individual must meet one of the following subgroup inclusion criteria to participate in this study.

SBMA subgroup:

1. Male
2. Genetically confirmed SBMA
3. Able to travel to the NIH
4. Greater than 18 years old

SBMA carriers:

1. Female
2. Genetically confirmed SBMA heterozygote
3. Able to travel to the NIH
4. Greater than 18 years old

Other motor neuron disease patients:

1. Diagnosis of motor neuron disease other than SBMA (e.g.. amyotrophic lateral sclerosis (ALS), spinal muscular atrophy)
2. Able to travel to the NIH
3. Greater than 18 years old
4. . Male

Healthy male control:

1. Male
2. No history or diagnosis of liver disease
3. No history of SBMA or other motor neuron disease
4. Greater than 18 years old
5. No diagnosis of diabetes or insulin resistance
6. No history of alcohol abuse within the last 1 year
7. No history of hyperlipidemia (LDL < 195) or hypertriglyceridemia (TAG < 225)

Healthy female control:

1. Female
2. No history or diagnosis of liver disease
3. No history of SBMA or other motor neuron disease
4. Greater than 18 years old
5. No diagnosis of diabetes or insulin resistance
6. No history of alcohol abuse within the last 1 year
7. No history of hyperlipidemia (LDL < 195) or hypertriglyceridemia (TAG < 225)

EXCLUSION CRITERIA:

* Diagnosed with an acquired or inherited liver disease eg., hepatitis B, hepatitis C, HIV, autoimmune hepatitis, cholestatic liver disease, Wilson s disease, iron overload disease, alpha-1 antitrypsin deficiency, hepatocellular carcinoma, (hepatic neoplasm or metastasis, etc.) or injury except for fatty liver disease.
* Contraindications to MRI such as a contraindicated non-removable metal device (i.e. pacemaker, defibrillator, insulin pump, metal clips, non-removable jewelry) or claustrophobia.
* Currently pregnant or pregnant within the past 6 months. Pregnant women are excluded from the study because of the known associated abnormalities in liver function that can occur in this population. The long term effects of MRI on the developing fetus are unknown and would present a risk with participation.

In addition to the above criteria, the patients receiving a liver biopsy will need to meet the additional exclusion criteria below:

* Coagulopathy (PT/PTT values that are prolonged >= 3 seconds from the upper limit of normal, including treatment with oral and parenteral anticoagulants), thrombocytopenia (< 70,000), abnormal bleeding time or platelet dysfunction.
* Taking anti-platelet agents for cardiovascular protection that cannot be safely stopped for the performance of the liver biopsy.
* Obesity, which is defined as a BMI>30 at the screenig visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to enroll men with genetically confirmed SBMA, age-matched healthy control men, SBMA carrier women, age-matched healthy control women and males with other motor neuron disease patients as disease controls.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Liver fat deposition measured by liver MRS proton density fat fraction at the site of the dome of the liver | Initial Visit and annual follow- up visits
  The primary outcome measures will be the liver fat deposition measured by liver MRS proton density fat fraction at the site of the dome of the liver. These measures will help us evaluate the prevalence and severity of fatty liver infiltration in SBMA patients compared to healthy controls.

SECONDARY OUTCOMES:
Assessment of liver injury by biochemical analysis and thephysiological measures | Initial Visit and annual follow-up visits
  The secondary outcome will be assessment of liver injury by biochemical analysis and the physiological measures (BMI, Free Testosterone, Total Testosterone). These outcome measures will help to evaluate whether the evaluated subjects have impairment of liver function by blood testing and other measurements. In addition, we hope to gain a better understanding of the relationship between testosterone levels and liver fat deposition.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Grunseich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Johnson B, Kokkinis A, Gai N, Shamim EA, Blackstone C, Fischbeck KH, Grunseich C. Nonalcoholic Fatty Liver Disease in Patients with Inherited and Sporadic Motor Neuron Degeneration. Genes (Basel). 2022 May 24;13(6):936. doi: 10.3390/genes13060936. PMID 35741698
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-N-0099.html